CLINICAL TRIAL: NCT02876601
Title: Defibrotide in the Human Endotoxemia Model -- an Exploratory Trial Investigating the Effects and the Mechanisms of Defibrotide
Brief Title: Defibrotide in the Human Endotoxemia Model --- an Exploratory Trial Investigating the Effects and the Mechanisms of Defibrotide
Acronym: LPS_DF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bernd Jilma (Other)
Responsible Party: Sponsor-Investigator, Bernd Jilma, Ao.Univ.Prof.Dr.med, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: LPS_DF Version 1.4
Record Dates: First submitted 2016-06-27; First posted 2016-08-24 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteers; Endotoxemia
Keywords: Coagulation; Inflammation; Defibrotide; Fibrinolysis
MeSH Terms: conditions — Endotoxemia; Thrombosis; Inflammation | interventions — defibrotide; Sodium Chloride; Lipopolysaccharides

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive LPS (n=16) or placebo (n=4) first. In each group they will undergo two study periods (crossover trial): a placebo period and a defibrotide period. The placebo group (n=4) will only be analyzed descriptively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Defibrotide/LPS (Active Comparator): 2ng/kg lipopolysaccharide period I: 6.25mg/kg bodyweight defibrotide or placebo (0.9% sodium chloride) period II: vice versa
  16 healthy volunteers will receive 2ng/kg bodyweight LPS plus Defibrotide or Placebo 4 healthy volunteers will receive 0.9% saline (NO LPS) plus Defibrotide or Placebo
  Interventions: Drug: Defibrotide; Drug: Lipopolysaccharide
- Placebo/LPS (Placebo Comparator): 2ng/kg lipopolysaccharide period I: 6.25mg/kg bodyweight defibrotide or placebo (0.9% sodium chloride) period II: vice versa
  16 healthy volunteers will receive 2ng/kg bodyweight LPS plus Defibrotide or Placebo 4 healthy volunteers will receive 0.9% saline (NO LPS) plus Defibrotide or Placebo
  Interventions: Drug: Placebo (0.9% sodium chloride); Drug: Lipopolysaccharide
- Defibrotide/Placebo (Other): Placebo (0.9% sodium chloride) period I: 6.25mg/kg bodyweight defibrotide or placebo (0.9% sodium chloride) period II: vice versa
  16 healthy volunteers will receive 2ng/kg bodyweight LPS plus Defibrotide or Placebo 4 healthy volunteers will receive 0.9% saline (NO LPS) plus Defibrotide or Placebo
  Interventions: Drug: Defibrotide; Drug: Placebo (0.9% sodium chloride bolus)
- Placebo/Placebo (Other): Placebo (0.9% sodium chloride) period I: 6.25mg/kg bodyweight defibrotide or placebo (0.9% sodium chloride) period II: vice versa
  16 healthy volunteers will receive 2ng/kg bodyweight LPS plus Defibrotide or Placebo 4 healthy volunteers will receive 0.9% saline (NO LPS) plus Defibrotide or Placebo
  Interventions: Drug: Placebo (0.9% sodium chloride); Drug: Placebo (0.9% sodium chloride bolus)

INTERVENTIONS:
Drug: Defibrotide — 6.25mg/kg bodyweight over 2h infusion
  Arms: Defibrotide/LPS; Defibrotide/Placebo
Drug: Placebo (0.9% sodium chloride) — (0.9% sodium chloride) infusion over 2h infusion
  Arms: Placebo/LPS; Placebo/Placebo
Drug: Lipopolysaccharide — bolus infusion of 2ng/kg bodyweight lps
  Arms: Defibrotide/LPS; Placebo/LPS
Drug: Placebo (0.9% sodium chloride bolus) — (0.9% sodium chloride) bolus infusion
  Arms: Defibrotide/Placebo; Placebo/Placebo

SUMMARY:
Defibrotide is an anti-inflammatory and anti-coagulatory agent approved for treatment of veno-occlusive disease. Although it has been in clinical use for almost 30 years, the exact mechanism of action has never been fully elucidated. Thus, the effects of defibrotide will be investigated in the human endotoxemia model in order to gather further information on its actions.

DETAILED DESCRIPTION:
Defibrotide (DF) is a highly complex polydisperse mixture of single-stranded phosphodiester oligodeoxyribonucleotides derived from the controlled depolymerization of porcine intestinal mucosal DNA. The entire mode of action remains unknown. Its actions may be summarized to pro-fibrinolytic, anti-inflammatory and anti-coagulatory actions. To better define the mechanisms of Defibrotide the effects of the substance will be investigated in the well-established endotoxemia model. Sixteen healthy volunteers will be randomized to receive LPS±defibrotide/placebo and four subjects will be randomized to receive Placebo± defibrotide/placebo in a single center, randomized, double blind, placebo controlled, two-way crossover trial. Immediately after a 2h infusion of 6,25mg/kg bodyweight defibrotide or placebo a LPS bolus of 2ng/kg bodyweight will be infused. Analyses will be performed by blood sampling at pre-defined time-points.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* <90kg body weight
* Normal findings in medical history and physical examination unless the investigator considers the abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers abnormalities to be clinically irrelevant
* Ability to understand the purpose and nature of the study, as well as the associated risks

Exclusion Criteria:

* Intake of any drugs that may interfere with the trial's endpoints or drugs (i.e. platelet inhibitors, anticoagulants, etc.)
* Positive results of HIV or hepatitis virology
* Acute illness with systemic inflammatory reactions
* Known allergies, hypersensitivities or intolerances to any of the used substances
* Acute or recent bleeding episodes, increased risk of bleeding at the discretion of the investigator
* Participation in an LPS trial within 6 weeks of the first study day
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Jilma, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be published in a peer-reviewed medical journal, individual data will not be presented or published, but may be made available by direct request to the PI (data may be made available in an anonymized fashion)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a crossover study. Of 20 healthy volunteers 16 were randomly assigned to receive LPS, while 4 received Placebo only. All participants underwent two study periods: A defibrotide and a placebo period.
  The system will not let us enter this study design of a crossover study. Only 20 healthy volunteers participated.
Groups:
- LPS+ First Defibrotide, Then Placebo: First Intervention:
  LPS: 2ng/kg bodyweight Defibrotide: 6.25mg/kg bodyweight over 2h infusion
  Washout for 6 weeks:
  Second Intervention:
  LPS: 2ng/kg bodyweight Placebo: 0.9% sodium chloride infusion over 2h infusion
- LPS+ First Placebo, Then Defibrotide: First Intervention:
  LPS: 2ng/kg bodyweight Placebo: 0.9% sodium chloride infusion over 2h infusion
  Washout for 6 weeks:
  Second Intervention:
  LPS: 2ng/kg bodyweight Defibrotide: 6.25mg/kg bodyweight over 2h infusion
- Placebo+ First Defibrotide, Then Placebo: 4 healthy volunteers were randomized not to receive LPS. However, they still received Placebo or Defibrotide. This group was included as another control group and to investigate the effects of Defibrotide in vivo.
  First Intervention:
  Placebo: bolus infusion of 0.9% sodium chloride solution Defibrotide: 6.25mg/kg bodyweight Defibrotide over 2 hours
  Washout: 6 weeks
  Second Intervention:
  Placebo: bolus infusion of 0.9% sodium chloride solution Placebo: 0.9% sodium chloride solution infusion over 2h
- Placebo+ First Placebo, Then Defibrotide: 4 healthy volunteers were randomized not to receive LPS. However, they still received Placebo or Defibrotide. This group was included as another control group and to investigate the effects of Defibrotide in vivo.
  4 healthy volunteers were randomized not to receive LPS. However, they still received Placebo or Defibrotide. This group was included as another control group and to investigate the effects of Defibrotide in vivo.
  First Intervention:
  Placebo: bolus infusion of 0.9% sodium chloride solution Placebo: 0.9% sodium chloride solution infusion over 2h
  Washout: 6 weeks
  Second Intervention:
  Placebo: bolus infusion of 0.9% sodium chloride solution Defibrotide: 6.25mg/kg bodyweight Defibrotide over 2 hours
Period: First Intervention (24 Hours)
Arm/Group | LPS+ First Defibrotide, Then Placebo | LPS+ First Placebo, Then Defibrotide | Placebo+ First Defibrotide, Then Placebo | Placebo+ First Placebo, Then Defibrotide
Started | 8 | 8 | 2 | 2
Completed | 8 | 8 | 2 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Washout (Minimum of 6 Weeks)
Arm/Group | LPS+ First Defibrotide, Then Placebo | LPS+ First Placebo, Then Defibrotide | Placebo+ First Defibrotide, Then Placebo | Placebo+ First Placebo, Then Defibrotide
Started | 8 | 8 | 2 | 2
Completed | 8 | 8 | 1 | 2
Not Completed | 0 | 0 | 1 | 0
Not completed — unforeseen unavailability | 0 | 0 | 1 | 0
Period: Second Intervention (24 Hours)
Arm/Group | LPS+ First Defibrotide, Then Placebo | LPS+ First Placebo, Then Defibrotide | Placebo+ First Defibrotide, Then Placebo | Placebo+ First Placebo, Then Defibrotide
Started | 8 | 8 | 1 | 2
Completed | 8 | 8 | 1 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LPS+ First Defibrotide, Then Placebo | LPS+ First Placebo, Then Defibrotide | Placebo+ First Defibrotide, Then Placebo | Placebo+ First Placebo, Then Defibrotide | Total
Number analyzed (Participants) | 8 | 8 | 2 | 2 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 2 | 2 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (9) | 29 (7) | 41 (8) | 21 (0) | 31 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 2
  Male | 8 | 8 | 2 | 0 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 8 | 8 | 2 | 2 | 20

OUTCOME MEASURES:

1. Primary Outcome: Prothrombin Fragments f1+2
Description: Based on the changes from baseline an area-under the concentration-time curve will be calculated and will be compared between the placebo and the verum phase within each subject. The respective arbitrary unit therefore is fold*h.
  The "placebo period" (4 subjects who did not receive lipopolysaccharide) was only included for a descriptive comparison, but not for statistical comparison
Time Frame: The parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h.
Population: The main statistical comparison was done for all subjects receiving LPS (defibrotide vs. placebo).
  The "placebo period" (4 subjects who did not receive lipopolysaccharide) was only included for a descriptive comparison, but not for statistical comparison
Measure: Median (Inter-Quartile Range); unit: fold-change*h
Groups:
- LPS Plus Defibrotide; LPS Plus Placebo: Intervention: 6.25mg/kg bodyweight defibrotide plus 2ng/kg bodyweight LPS bolus infusion
- Placebo Plus Defibrotide: Intervention: placebo infusion (0.9% sodium chloride) plus 2ng/kg bodyweight LPS bolus infusion
- Placebo Plus Placebo: Intervention: placebo (0.9% sodium chloride) infusion placebo bolus infusion (0.9% sodium chloride)
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold-change*h | 31.1 [16.96 to 61.6] | 34.08 [20.38 to 60.8] | 27.41 [27.21 to 46.48] | 36.02 [23.64 to 51.95]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.408, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Thrombin-Antithrombin Complexes
Description: as for outcome 1
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Placebo: Intervention: placebo infusion (0.9% sodium chloride) plus 2ng/kg bodyweight LPS bolus infusion
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus placebo bolus infusion (0.9%sodium chloride)
- Placebo Plus Placebo: Intervention: placebo infusion (0.9% sodium chloride) plus placebo bolus infusion (0.9% sodium chloride)
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 23.39 [15.19 to 32.52] | 27.4 [21.47 to 41.57] | 17.46 [15.58 to 20.46] | 21.83 [16.09 to 23.26]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.148, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Plasmin-Antiplasmin Complexes
Description: as for outcome 1
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, and 6h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide and 2ng/kg bodyweight LPS bolus
- LPS/Placebo: Intervention: placebo infusion (0.9% sodium chloride) and 2ng/kg bodyweight LPS bolus
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide and Placebo bolus (0.9% sodium chloride)
- Placebo Plus Placebo: Intervention: placebo infusion (0.9% sodium chloride) and placebo bolus infusion (0.9% sodium chloride)
Arm/Group | LPS Plus Defibrotide | LPS/Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 11.8 [9.59 to 15.12] | 9.99 [8.15 to 13.16] | 7 [6.31 to 7.19] | 7.12 [6.34 to 7.79]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS/Placebo; Test type: Superiority; p = 0.039, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Tumor Necrosis Factor (TNF)-Alpha
Description: Based on the changes from baseline an area-under the concentration-time curve will be calculated and will be compared between the placebo and the verum phase within each subject.
  The respective arbitrary unit therefore is fold*h.
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: The "placebo period" (4 subjects who did not receive lipopolysaccharide) was only included for a descriptive comparison, but not for statistical comparison
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus 2ng/kg lipopolysaccharide bolus infusion
- LPS Plus Placebo: Intervention: 6.25mg/kg bodyweight defibrotide plus placebo bolus infusion (0.9% sodium chloride)
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus Placebo infusion (0.9% sodium chloride
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 286 [162 to 453] | 326 [172 to 366] | 28.08 [22.19 to 28.35] | 21.01 [16.75 to 25.27]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.642, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Tissue-type Plasminogen Activator
Description: as for outcome 4
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus 2ng/kg bodyweight lipopolysaccharide
- LPS Plus Placebo: Intervention: Placebo infusion (0.9% sodium chloride) plus 2ng/kg bodyweight LPS
- Placebo Plus Defibrotide: Intervention: placebo bolus (0.9% sodium chloride) plus 6.25mg/kg bodyweight defibrotide
- Placebo Plus Placebo: Intervention: placebo bolus (0.9% sodium chloride) plus placebo (0.9% sodium chloride) infusion
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 21.8 [14.9 to 29.3] | 17 [13.9 to 23.9] | 20.57 [19.75 to 21.45] | 23.54 [21.72 to 24.78]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.026, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Interleukin-6
Description: as for outcome 4
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus infusionbolus infusion of 2ng/kg bodyweight LPS
- LPS Plus Placebo: Intervention: Bolus infusion of 2ng/kg bodyweight LPS plus Placebo (0.9% sodium chloride)
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight Defibrotide infusion plus Placebo (0.9% sodium chloride)
- Placebo Plus Placebo: Intervention: Placebo (0.9% sodium chloride) bolus infusion plus placebo (0.9% sodium chloride) infusion
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 1543 [815 to 2919] | 1144 [22 to 1923] | 35 [32 to 113] | 31 [23 to 51]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.326, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: E-Selectin
Description: as for outcome 4
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: Defibrotide 6.25mg/kg infusion plus bolus infusion of 2ng/kg bodyweight LPS
- LPS Plus Placebo: Intervention: placebo (0.9% sodium chloride) infusion plus 2ng/kg bodyweight LPS bolus infusion
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide infusion plus placebo (0.9% sodium chloride) bolus infusion
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 35 [32 to 40] | 33 [24 to 45] | 21 [18 to 36] | 41 [20 to 63]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.796, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Plasminogen Activator Inhibitor 1
Description: as for outcome 4
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide infusion plus 2ng/kg LPS bolus infusion
- LPS Plus Placebo: Intervention: placebo (0.9% sodium chloride) infusion plus 2ng/kg bodyweight LPS
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide plus placebo (0.9% sodium chloride) infusion
- Placebo Plus Placebo: Intervention: placebo (0.9% sodium chloride) infusion plus placebo (0.9% sodium chloride) bolus infusion
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 216 [32 to 898] | 477 [49 to 1000] | 25 [25 to 29.5] | 24.86 [22.7 to 25]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.918, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Von Willebrand Factor Antigen
Description: Based on the changes from baseline an area-under the concentration-time curve will be calculated and will be compared between the placebo and the verum phase within each subject. The quantification of von Willebrand Factor is based on reference values and results are in % of "normal".
  The respective arbitrary unit therefore is %*h.
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: %*h
Groups:
- Placebo Plus Defibrotie: Intervention: 6.25mg/kg bodyweight defibrotide plus placebo bolus infusion (0.9% sodium chloride solution)
- Placebo Plus Placebo: Intervention: Placebo (0.9% sodium chloride solution) infusion plus placebo bolus infusion (0.9% sodium chloride)
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotie | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
%*h | 54 [41 to 70] | 53 [41 to 65] | 27 [27 to 31] | 26 [24 to 29]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.877, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Clotting Time in Thromboelastometry
Description: In this analysis, first of all a ratio of the measurement time point to the baseline was calculated. Thereafter deltas (baeline-ratio) were calculated. With the results an AUC was calculated.
  The respective arbitrary unit therefore is fold*h.
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h, 24h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight LPS plus bolus infusion of 2ng/kg bodyweight LPS
- LPS Plus Placebo: Intervention: placebo infusion (0.9% sodium chloride solution) plus bolus infusion of 2ng/kg bodyweight LPS
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight defibrotide infusion plus placebo (0.9% sodium chloride solution) bolus infusion
- Placebo Plus Placebo: Intervention: placebo (0.9%sodium chloride solution) infusion plus placebo bolus infusion (0.9% sodium chloride solution)
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 1.12 [0.8 to 1.43] | 1.12 [1.04 to 1.41] | -0.2 [-6 to 2.17] | 2.14 [0.31 to 4.28]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.423, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Maximum Lysis in Thromboelastometry
Description: as for outcome 4
Time Frame: This parameter was assessed at baseline, at 0h, 1h, 2h, 4h, 6h and AUC was calculated based on these measurements.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: fold*h
Groups:
- LPS Plus Defibrotide: Intervention: 6.25mg/kg bodyweight infusion plus 2ng/kg bodyweight LPS bolus infusion
- LPS Plus Placebo: Intervention: placebo infusion (0.9% sodium chloride infusion) plus 2ng/kg bodyweight LPS bolus infusion
- Placebo Plus Defibrotide: Intervention: 6.25mg/kg bodyweight infusion plus placebo (0.9% sodium chloride solution) bolus infusion
Arm/Group | LPS Plus Defibrotide | LPS Plus Placebo | Placebo Plus Defibrotide | Placebo Plus Placebo
Number analyzed (Participants) | 16 | 16 | 3 | 4
fold*h | 7.9 [7.1 to 10.1] | 7.7 [6.6 to 9] | 6.84 [6.72 to 7.07] | 6.85 [6.32 to 7.05]
Statistical Analysis 1: Comparison: LPS Plus Defibrotide vs LPS Plus Placebo; Test type: Superiority; p = 0.938, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: For the individual subject, adverse events were assessed during every study visit (screening, study day1, study day 2, follow up) during the whole study. The whole study period lastet for a minimum of 8 weeks, but could be longer for individual subjects (washout period was a minimum of 6 weeks). The respective time frame could therefore differ between the individual subjects but was a minimum of 8 weeks.
Groups:
- Defibrotide Plus LPS: Intervention: 6.25mg/kg bodyweight defibrotide infusion plus 2ng/kg bodyweight LPS infusion
- Placebo Plus LPS: Intervention: placebo infusion (0.9% sodium chloride solution) plus 2ng/kg bodyweight LPS infusion
- Defibrotide Plus Placebo: Intervention: 6.25mg/kg bodyweight defibrotide infusion plus placebo bolus infusion (0.9% sodium chloride solution)
- Placebo/Placebo: Intervention: placebo infusion (0.9% sodium chloride solution) plus placebo bolus infusion (0.9% sodium chloride solution)
Arm/Group | Defibrotide Plus LPS | Placebo Plus LPS | Defibrotide Plus Placebo | Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 13/16 | 15/16 | 1/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Defibrotide Plus LPS (N=16) | Placebo Plus LPS (N=16) | Defibrotide Plus Placebo (N=3) | Placebo/Placebo (N=4)
Headache (Nervous system disorders) | 13 (13) | 11 (11) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flu-like Symptoms (General disorders) | 6 (6) | 6 (6) | 0 (0) | 0 (0)
Arthralgia (General disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0) — Feeling Cold
Impaired Concentration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Precollapse (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urticarial rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT02876601/Prot_SAP_000.pdf